CLINICAL TRIAL: NCT05015283
Title: Efficacy and Safety of One-anastomosis Versus Roux-en-Y Gastric Bypass for Type 2 Diabetes Remission (ORDER): a Multi-centric, Randomized, Open-label, Superiority Trial
Brief Title: Efficacy and Safety of One-anastomosis Versus Roux-en-Y Gastric Bypass for Type 2 Diabetes Remission
Acronym: ORDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); The Third Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Soochow University (Other); The Third People's Hospital of Chengdu (Other); Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigator, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFH-ORDER
Record Dates: First submitted 2021-07-20; First posted 2021-08-20 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Type2 Diabetes; Complication of Bariatric Procedure
Keywords: Bariatric surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic One-anastomosis gastric bypass (Experimental): In this group, the bariatric procedure is laparoscopic one-anastomosis gastric bypass, all operations follow the same standard operating procedure.
  Interventions: Procedure: The laparoscopic One-anastomosis gastric bypass will consist of:
- Laparoscopic Roux-en-Y gastric bypass (Active Comparator): In this group, the bariatric procedure is laparoscopic Roux-en-Y gastric bypass, all operations follow the same standard operating procedure.
  Interventions: Procedure: The laparoscopic Roux-en-Y gastric bypass will consist of:

INTERVENTIONS:
Procedure: The laparoscopic One-anastomosis gastric bypass will consist of: — gastrointestinal anastomosis: anterior colon and posterior stomach gastrointestinal anastomosis size: diameter < 1.5cm, linear anastomosis length 2.5cm biliary and pancreatic branches 200cm, food branches 100cm exact relationship with mesangial defect
  Arms: Laparoscopic One-anastomosis gastric bypass
Procedure: The laparoscopic Roux-en-Y gastric bypass will consist of: — the laparoscopic Roux-en-Y gastric bypass gastric sac size < 30ml gastrointestinal anastomosis: anterior colon and posterior stomach gastrointestinal anastomosis size: diameter < 1.5cm, linear anastomosis length 2.5cm biliary and pancreatic branches 50cm, food branches 150cm exact relationship with mesangial defect
  Arms: Laparoscopic Roux-en-Y gastric bypass

SUMMARY:
Diabetes mellitus (T2DM) is the most common complication of obesity patients. According to previous literature reports, weight loss and metabolic surgery are powerful means to treat obesity complicated with T2DM. Roux-en-Y gastric bypass (RYGB) is the standard operation recommended by the international society. One-anastomosis gastric bypass (OAGB) was recommended by IFSO（the International Federation for the Surgery of OBESITY AND METABOLIC DISORDERS ） in 2018.

In this study, two kinds of metabolic surgery will be compared. At present, focusing on the above two operations, only two effective randomized controlled clinical studies have been carried out, among which one single-center clinical study has been followed up for 2 years, and the primary end point is weight loss; Another multicenter study, with a 2-year follow-up, showed that the primary end point was weight loss, and the secondary index was the effectiveness of two surgical methods in the treatment of T2DM.There is still a lack of evidence-based evidence for the effectiveness and safety of the two surgical methods in the treatment of T2DM. This study will make high-level evidence about the advantages and disadvantages of OAGB and RYGB in the treatment of T2DM.

In this study, a number of centers with rich experience and clinical research experience in weight loss and metabolic surgery in Asia will be combined to complete the enrollment of 248 patients. Those who meet the standards will be randomly divided into two kinds of operations, and they will be followed up for 5 years on schedule. The rate of lost follow-up is controlled within 20%, and the data integrity is controlled within 95%. Taking the blood glucose remission rate of type 2 diabetes as the main observation index, the prospective verification shows that OAGB is clinically effective in treating obesity with type 2 diabetes compared with RYGB.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old, Male/Female, East Asian population
* 50 kg/m2≥BMI≥27.5kg/m2
* Type 2 diabetes duration ≥6 months
* HbA1c≥7.0%
* Currently receiving one or more oral/injectable hypoglycemic drugs (insulin /glucagon-like peptide-1 receptor agonist)
* Recommendation for OAGB/RYGB evaluated by a multidisciplinary team

Exclusion Criteria:

* Underwent gastrointestinal surgery (gastric/duodenal surgery or bariatric surgery)
* Fasting C-peptide level lower than 1/2 normal minimum
* Active gastrointestinal ulcer is present
* Helicobacter pylori infection is present
* A history of serious cardiovascular and cerebrovascular diseases (myocardial infarction, stroke, etc.)
* A history of cirrhosis (Child-Pugh≥A)
* A history of chronic kidney disease (eGFR )< 60 ml/min / 1.73 m2)
* Inflammatory bowel disease is present (ulcerative colitis, Crohn's disease)
* Chronic anemia is present, Hgb for male <100g/L, for female <90g/L
* A desire to conception during the study period
* Uncontrolled mental and psychological disorders are present
* Expected survival<5 years of end-stage disease or previous/current malignant tumor
* Participated in clinical studies/trials that have the conflict of interest with the study
* Unable to understand, refuse to participate and sign the informed consent
* Gallstones require cholecystectomy
* Reflux esophagitis above grade A

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
One year after operation, the complete remission rate of type 2 diabetes mellitus [HbA1c < 6%, fasting plasma glucose < 5.6 mmol/L, no need to use any hypoglycemic drugs] | 1 year after surgery
  Complete remission of type 2 diabetes mellitus: the blood sugar HbA1c<6.0% and fasting plasma glucose< 5.6 mmol/L can be controlled only by changing lifestyle intervention without taking hypoglycemic agents after operation. Partial remission: blood glucose can be controlled only by changing lifestyle intervention after operation. HbA1c<6.5%, fasting plasma glucose 5.6~6.9mmol/L, and blood glucose 7.8~11.0mmol/L 2 hours after meal. Failure: blood sugar was relieved once, and then returned to the preoperative level.Unified OGTT measurement method

SECONDARY OUTCOMES:
The remission rate of type 2 diabetes mellitus | 5 years after surgery
  [HbA1c < 6%, with or without hypoglycemic drugs] Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
The change of HbA1c | 5 years after surgery
  Changes of glycosylated hemoglobin (HbA1c) compared with baseline.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
HbA1c value | 5 years after surgery
  The value of HbA1c.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
The change of fasting blood glucose | 5 years after surgery
  Changes of fasting blood glucose compared with baseline.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Fasting blood glucose level | 5 years after surgery
  The fasting blood glucose level.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Fasting plasma insulin | 5 years after surgery
  The value of fasting plasma insulin.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Diabetes medication | 5 years after surgery
  Follow up was used to observe whether the dosage of postoperative diabetes was reduced.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Fasting blood lipids | 5 years after surgery
  The value of fasting blood lipids.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Changes of arterial blood pressure (SBP, DBP) | 5 years after surgery
  The change of arterial blood pressure (SBP, DBP).Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
The excess weight loss (%EWL) and the total weight loss (%TWL) after surgery. | 5 years after surgery
  %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2),%TWL=[(initial weight)-(post-op weight)]/initial weight.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Change waist circumference (cm) according to absolute waist circumference | 5 years after surgery
  Change waist circumference (cm) according to absolute waist circumference.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Incidence of medical and surgical complications | 5 years after surgery
  Incidence of medical and surgical complications (anastomotic leakage, bile reflux, intestinal obstruction, anastomotic ulcer, anastomotic stenosis, internal hernia, chronic gastritis, esophagitis, iron deficiency anemia ...) Visit 1:Post-op 1 month (+7 Days) Visit 2: Post-op 3 months(+7 Days) Visit 3: Post-op 6 months(14 Days) Visit 4: Post-op 12 months (+30 Days) Visit 5：Post-op 24 months (±30 Days) Visit 6:Post-op 36 months (±30 Days) Visit 7：Post-op 60 months (±30 Days)
Incidence of surgical complications | 5 years after surgery
  According to the grade of surgical complications, proportion of surgical complications in the total number.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Surgery time | Surgery day (day 0) record
  Surgery time.Visit 1: Surgery day (day 0) record
Average length of stay, based on the length of stay from operation (surgery day =day0) to the end of hospitalization | 30 days after surgery
  Average length of stay, based on the length of stay from operation (surgery day =day0) to the end of hospitalization.Visit 1: Surgery day (day 0) record
Postoperative quality of life of patients, according to Impact Weight Quality Of Life questionnaire for weight loss surgery, scores were obtained | One day before surgery,5 years after surgery
  According to Impact Weight Quality Of Life questionnaire for weight loss surgery, scores were obtained.The higher the score, the better the quality of life. Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Postoperative gastroesophageal reflux | One day before surgery,5 years after surgery
  Evaluate according to gastroesophageal reflux disease questionnaire. The higher the score, the more likely there is gastroesophageal reflux. Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Diarrhea frequency | One day before surgery,5 years after surgery
  Based on gastrointestinal symptom rating scale.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)
Dumping syndrome and hypoglycemia symptoms | 5 years after surgery
  Dumping syndrome and hypoglycemia symptoms.Dumping syndrome and hypoglycemia symptoms will be evaluated by questionnaire.Visit 1: Baseline Visit (Day 0-1) Visit 2:Post-op 1 month (+7 Days) Visit 3: Post-op 3 months(+7 Days) Visit 4: Post-op 6 months(14 Days) Visit 5: Post-op 12 months (+30 Days) Visit 6：Post-op 24 months (±30 Days) Visit 7:Post-op 36 months (±30 Days) Visit 8：Post-op 60 months (±30 Days)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, M.D.;Ph.D, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
1. Will individual deidentified participant data (including data dictionaries) will be shared: Yes
  2. what data in particular will be shared: Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
  3. what other documents will be available: study portocol
  4. when will data be availuble (start and end dates): Beginning 6 months and ending 24 months following article publicaiton.
  5. With whom: Investigators whose proposed use of the data has been approved by an independent review commmittee identified for this purepose.
  6. For what types of analysis: For individual participant data meta-analysis.
  7. By what mmechanism will data be made available: Proposals should be directed to zhangzht@ccmu.edu.cn to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 24 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Derived] Li M, Liu Y, Lee WJ, Shikora SA, Robert M, Wang W, Wong SKH, Kong Y, Tong DKH, Tan CH, Zeng N, Zhu S, Wang C, Zhang P, Gu Y, Bai R, Meng F, Mao Z, Zhao X, Wu L, Liu Y, Zhang S, Zhang P, Zhang Z. Efficacy and safety of one anastomosis gastric bypass versus Roux-en-Y gastric bypass for type 2 diabetes remission (ORDER): protocol of a multicentre, randomised controlled, open-label, superiority trial. BMJ Open. 2022 Sep 29;12(9):e062206. doi: 10.1136/bmjopen-2022-062206. PMID 36175102